CLINICAL TRIAL: NCT01644578
Title: Prospective Use of Real-time MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-005887
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2019-06

CONDITIONS: Evaluate the Role of Real-time Imaging in Needle Placement; Evaluate the Workflow and Effectiveness of Realtime Imaging Versus Standard MR Imaging
Keywords: MRI; real-time imaging; workflow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Real-time imaging for MRI-guided procedures (Other): Real-time imaging for improvement of workflow in MRI-guided procedures
  Interventions: Procedure: Real-time imaging for MRI-guided procedures

INTERVENTIONS:
Procedure: Real-time imaging for MRI-guided procedures — Real-time imaging for improvement of workflow in MRI-guided procedures

SUMMARY:
This research study is being done to look at a new MRI imaging software, Siemens Interventional Software, to see if we can improve our ability to see and treat cancerous tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a percutaneous MR guided procedure

Exclusion Criteria:

* Pregnant Women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-10; Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Determine the time required for each step for needle placement | Intra-procedure

SECONDARY OUTCOMES:
Determine ease of use of the software | Intra-procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Woodrum, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials